CLINICAL TRIAL: NCT05289102
Title: An Extended Postnatal Program: a Randomized Controlled Trial
Brief Title: The Value of an Extended Postnatal Program.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Protocol ID:277301
Record Dates: First submitted 2022-02-08; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-02

CONDITIONS: Postpartum
Keywords: Postpartum period; Breast Feeding; Gynaecology; Birth; Contraception
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: This is a non-blind, two-arm randomized controlled multi-center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two postpartum visits. (Experimental): Group 1 serves as an intervention group (experimental). All enrolled women in the intervention group were in connection with the inclusion given two pre-booked postpartum care visits. One early at 3 weeks postpartum, and one later at 7 weeks postpartum.
  Interventions: Other: One postpartum visit.
- One postpartum visit. (Active Comparator): Group 2 serves as a control group (active comparator). All enrolled women in the control group were in connection with the inclusion given one pre-booked postpartum care visit at 7 weeks postpartum according to the traditional postpartum care.
  Interventions: Other: Two postpartum visits.

INTERVENTIONS:
Other: Two postpartum visits. — Group 1 serves as an intervention group (experimental). All enrolled women in the intervention group were in connection with the inclusion given two pre-booked postpartum care visits. One early at 3 weeks and one later at 7 weeks postpartum.
  Arms: One postpartum visit.
Other: One postpartum visit. — Group 2 serves as a control group (active comparator). All enrolled women in the control group were in connection with the inclusion given one pre-booked postpartum care visit at 7 weeks postpartum according to the traditional postpartum care.
  Arms: Two postpartum visits.

SUMMARY:
The objective was to study and evaluate earlier and extended postpartum care visits (week 3 and 7) compared to the current structure of one traditional visit 7 weeks postpartum.

In Sweden there is an organized system of antenatal and postnatal care based on local maternity clinics that are run by midwives who collaborate with obstetricians and surrounding hospitals. Pregnant women are regularly assessed by a midwife during their antenatal care. If complications occur, they are assessed by an obstetrician at the maternity clinic or at the nearest hospital. Postnatally a follow up visit to the same maternity clinic is offered usually about 6-12 weeks postpartum. Nowadays a healthy primigravid woman with a full-term pregnancy and a healthy child leaves the hospital within 6-24 hours postpartum. Many women experience the time between leaving the hospital until the postnatal follow up visit as too long. It is described that women missing early feedback regarding the experience of giving birth, breastfeeding, the transition of parenthood and sometimes physical examination.The eligible women enrolled were asked if they wanted to voluntarily participate in the trial about postpartum care.The women participating were recruited in pregnancy week 37 and offered to join, and if interested randomly divided into one of two groups. One control group who received a traditional postpartum care visit, that is one visit to a midwife 7 weeks postpartum, and one intervention group where the participating women were invited to two visits to the midwife; 3 weeks postpartum and then an additional visit 7 weeks postpartum. At the end of the visits both in the intervention group and in the control group the women completed a questionnaire given them via a Quick Response-code (QR-code) to fill in on their mobile phone. The questionnaire contained questions regarding delivery, breastfeeding, satisfaction with recieved care, evaluation of postpartum care offered, satisfaction with the visit and birth control.

The hypothesis is that two visits (week 3 and 7) will have an impact on womens health, wellbeing, satisfaction and contraceptive use postpartum.

DETAILED DESCRIPTION:
Trial Design and Setting. This is a non-blind, two-arm randomized controlled multi-center trial taking place in six different maternity clinics in Gothenburg and Molndal, Sweden (maternity clinics Frolunda Torg, Molndal, Gibraltargatan, Linné, Gamlestan, Angered).

Enrollment was conducted between January 2019 and February 2020. Pregnant women attending prenatal care in one of the included maternity clinics were approached.The women participating were recruited in pregnancy week 37 and offered to join, and if interested randomly divided into one of two groups The information about the trial was given in written and orally. The eligible women also had the opportunity to ask further questions to their pregnancy caregiver and patient responsible midwife. The information comprised that the participants was not given any merits or demerits if participating, decline or withdraw during the study. Eligible women who agreed to participate then gave written informed consent to the study. The randomization occurred after eligibility and consent.

Participants were randomly assigned to one of the trial groups, intervention, or control group. The randomization procedure was compiled together with a statistician. The chosen randomization procedure was based on the participants date of birth. If the participant was born on an even date of birth, she was allocated to intervention group. If the participant had an uneven date of birth, she was allocated to the control group. No co-location or stratification used.

Intervention and control. All enrolled women in the intervention group were in connection with the inclusion given two pre-booked postpartum care visits, one early at 3 weeks postpartum, and one later at 7 weeks postpartum. The control group received one pre-booked appointment at 7 weeks postpartum according to the traditional care.

At the first visit after giving birth the participants in the intervention group (3 week) as well as in the control group (7 week) were given opportunity to discuss breastfeeding, birth relating questions, and help with potential gynaecological problems such as ruptures and bleeding. The women were also given information regarding fertility postpartum and offered contraceptive counseling. The second visit (7 week) out of two in the intervention group gave opportunity to follow up the first 3 week visit. In connection to all visits the participants received a questionnaire via QR-code to fill in on the participants mobile phone/or as a paper questionnaire.

Data Collection. All participants in the intervention group or in the control group filled in the questionnaire through their phone/paper questionnaire close to their visit at the antenatal clinic . To ensure confidentiality all participants received an individual 4-digit code to use when answering the questionnaires. The code key is kept only for research responsible. The source data were collected using the esMaker, a secure web-based design for surveys. The data containing information on baseline characteristics such as nationality, age, BMI, height, weight, method of birth and parity. Questions regarding satisfaction with received care, whether fully-lactating, non-lactating, part lactating. Also questions regarding the participants opinion/satisfaction on the number of visits they received in the study, if they would have wished fewer/additional/latter/prior visits in relation the time of giving birth.

The questionnaires also comprise questions regarding contraceptive use, method of contraception and timing for start of contraceptive use postpartum.

One year after delivery the women in both the intervention group and the control group had a follow-up questionnaire.

Sample Size. Calculated sample size of a minimum of (n=400) in each group to achieve 80% power at a significance level at 0.05 and to detect a 10% difference between the independent groups (intervention and control group). A p-value <.05 was considered statistically significant.

Statistical Methods. Statistical analysis was performed using Statistical Analysis System (SAS) version 9.4 following a predetermined statistical analysis plan. Initial analyses assessed for the equivalency of study groups on baseline characteristics using Mantel-Haenszel Chi Square tests to compare proportions for categorical variables and Fisher exact test to compare means for continuous variables. Risk ratios and 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Attending patient for prenatal care at one of the included maternal clinics,
* During the recruitment period was in the 37th pregnancy week,
* Independent and fluent in English or Swedish

Exclusion Criteria:

* Age >18.
* Not fluent in English or Swedish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — A woman who deliver a child close to enrolment
Enrollment: 1159 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2021-03-28 (Actual)

PRIMARY OUTCOMES:
Satisfaction with visit after having two visits. | 7 weeks after delivery.
  In the intervention group; Satisfaction differences will be measured by using a five-grade scale where 1 stand for "Strongly disagree" and 5 Stands for "Strongly agree" in the questionnaire.
Satisfaction with visit after having one visit. | 7 weeks after delivery.
  In the control group; Satisfaction differences will be measured by using a five-grade scale where 1 stand for "Strongly disagree" and 5 Stands for "Strongly agree" in the questionnaire.
Breastfeeding after having two visits. | 7 weeks after delivery
  In the intervention group;Change in lactating measured by questionnaires. The participants were asked to report their breastfeeding. The answering alternatives werefully-lactating, non-lactating and part lactating.
Breastfeeding after having one visit. | 7 weeks after delivery
  In the control group;Change in lactating measured by questionnaires. The participants were asked to report their breastfeeding. The answering alternatives werefully-lactating, non-lactating and part lactating.
Breastfeeding continued in month for the intervention group. | 1 year after delivery.
  Lactating at one year follow-up vill be measured by a questionnaire for all participating women one year after delivery. Participants were asked to report if the were still breastfeeding or if stopped breastfeeding for how many month since delivery.
Breastfeeding continued in month for the control group. | 1 year after delivery.
  Lactating at one year follow-up vill be measured by a questionnaire for all participating women one year after delivery. Participants were asked to report if the were still breastfeeding or if stopped breastfeeding for how many month since delivery.
Opinion on the number and content of the visit after having two visits. | At 7 weeks after delivery.
  Intervention group;The women were asked in the questionnaire to report if they were satisfied. The answering alternatives were "It is enough with one visit" "I would preferred to have two visits close to the delivery and one a little bit later" . For you who got one visit 7 weeks pospartum what had you preferred to talk about if you had a visit 3 weeks after delivery? (You may choose more than one alternative)? 1. The delivery 2. Breastfeeding 3. Gyneacological problems, 4.contraception 5. Other emergent problems after delivery.
Opinion on the number and content of the visit after having one visit. | At 7 weeks after delivery.
  Control group;The women were asked in the questionnaire to report if they were satisfied. The answering alternatives were "It is enough with one visit" "I would preferred to have two visits close to the delivery and one a little bit later" . For you who got one visit 7 weeks pospartum what had you preferred to talk about if you had a visit 3 weeks after delivery? (You may choose more than one alternative)? 1. The delivery 2. Breastfeeding 3. Gyneacological problems, 4.contraception 5. Other emergent problems after delivery.
Contraceptive use after having two visits. | 7 weeks postpartum
  Intervention group; Change in contraception use measured by a questionnaire. The questonnaire contains questions to answer regarding 1. prevalence of contraception, 2. contraceptive method used and 3. time for start of contraception
Contraceptive use after having one visit. | 7 weeks postpartum
  Control group; Change in contraception use measured by a questionnaire. The questonnaire contains questions to answer regarding 1. prevalence of contraception, 2. contraceptive method used and 3. time for start of contraception
Contraceptive use and compliance with method used after having two visits. | 1 year after delivery
  Intervention group;The participated women were asked about change in contraception method and pregnancies during the first year after delivery. The answering alternatives were 1. do you still use the same contraceptive method? 2. If not what method have you changed to? 3. Why did you changed or stopped using the method? 4. Have you been pregnant? 5. Are you pregnant now?
Contraceptive use and compliance with method used after having one visit. | 1 year after delivery
  Control group;The participated women were asked about change in contraception method and pregnancies during the first year after delivery. The answering alternatives were 1. do you still use the same contraceptive method? 2. If not what method have you changed to? 3. Why did you changed or stopped using the method? 4. Have you been pregnant? 5. Are you pregnant now?
Seeking medical care postpartum after having two visits. | 1 year after delivery.
  Intervention group; Seeking medical care the first three month postpartum measured by the questionnaire one year after delivery. The women were asked to report if they had been seeking medical care and if answer Yes on this question they could report reason.
Seeking medical care postpartum after having one visit. | 1 year after delivery.
  Control group; Seeking medical care the first three month post partum measured by the questionnaire one year after delivery. The women were asked to report if they had been seeking medical care and if answer Yes on this question they could report reason.

CONTACTS AND LOCATIONS:
Overall Officials: Ingela Lindh, PhD, Principal Investigator — Department of Obstetrics and Gynaecology, Sahlgrenska University Hospital, Sweden
Locations (1):
- Ingela Lindh, Västra Frölunda, Sweden

IPD SHARING:
Plan to Share IPD: No